CLINICAL TRIAL: NCT05187897
Title: CHV-NEO: Community-based Digital Communication to Support Neonatal Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); BRAC University (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Keshet Ronen, Assistant Professor, School of Public Health: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00012725; R01HD103581 (NIH)
Record Dates: First submitted 2021-12-24; First posted 2022-01-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Death; Perinatal Death
Keywords: SMS; Essential Newborn Care; Kenya; Community Health Volunteer; Neonate; mHealth; Implementation Science
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: Facilities will be randomized to 1) Interactive two-way SMS dialogue integrated into CHV workflow or 2) Control (standard care), using 1:1 allocation. All participants at each study facility will receive the assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Control (No Intervention): CHVs based at facilities in the control arm will continue to implement the standard of care.
- CHV-NEO Intervention (Experimental): CHVs based at facilities in the Intervention arm will implement the integrated CHV-NEO two-way SMS messaging intervention with their clients.
  Interventions: Behavioral: CHV-NEO

INTERVENTIONS:
Behavioral: CHV-NEO — CHV-NEO is a two-way SMS platform that supports communication between mothers and community health volunteers between home visits. The platform engages mothers with SMS communication and brings timely information and support - asking critical questions at crucial times in order to assess the needs and health of newborns and assist in care seeking decisions. The CHV-NEO SMS intervention is integrated into the current digital community health toolkit (dCHT) to support CHV workflow.
  Arms: CHV-NEO Intervention

SUMMARY:
Neonatal mortality (defined as death in the first 28 days of life) remains unacceptably high in sub-Sarahan Africa. The concentrated risk of neonatal illness in the first weeks of life and its potential to rapidly deteriorate means that expanding mothers' access to timely information and support during this period is critical to reducing neonatal mortality. This cluster-randomized control trial aims to integrate a 2 way interactive SMS text messaging intervention into existing digital infrastructure supporting Community Health Volunteer (CHV) workflow in Western Kenya (dCHT) to enable remote communication by mothers with CHVs between home visits.

DETAILED DESCRIPTION:
In Kenya, the neonatal mortality rate is 22.6 per 1000 live births, ranking among the countries with the highest number of neonatal deaths (~40,000 per year). Community health volunteers (CHVs) are a large cadre of lay health workers whose role is to promote access to preventative care and treatment in resource-limited settings. In Kenya, CHVs conduct monthly home visits to pregnant and postpartum women to provide education and screen for complications. Several counties in Kenya have adopted a digital community health toolkit (dCHT) that supports CHV workflow by tracking clients, managing tasks, and guiding home visits. Even so, the concentrated risk of neonatal illness in the first weeks of life and its potential to rapidly deteriorate mean that even monthly home visits leave mothers and neonates in need of on-demand support.

Our team developed an interactive SMS text messaging intervention, Mobile WACh Neo (NEO), that connects mothers with healthcare workers remotely in the high-risk period immediately following birth to improve maternal and neonatal health. NEO sends automated, theory-based, actionable daily messages that systematically guide mothers to evaluate neonatal danger signs, and facilitates real-time dialogue with a healthcare worker to triage medical concerns and augment maternal social support.

The overarching goal of this project is to integrate NEO interactive SMS into the existing digital infrastructure supporting CHV workflow in Western Kenya (dCHT) to enable remote communication by mothers with CHVs between home visits. This is a cluster-randomized control trial consisting of 20 facility clusters (10 control, 10 intervention) in Western Kenya.

AIM 1: Employ a human-centered design approach to develop a NEO interactive SMS module in the dCHT, named CHV-NEO.

AIM 2: a) Evaluate CHV-NEO's impact on neonatal mortality, b) clinic visit attendance, and caregiver provision of essential newborn care (cord care, thermal care and initiation of breastfeeding), in a pragmatic cluster-randomized trial.

AIM 3: a) Determine the effect of CHV-NEO on CHV and supervisor workflow, and b) evaluate determinants of CHV-NEO's acceptability, adoption and fidelity of use.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 26-36 weeks gestation
* Daily access to a mobile phone (own or shared)
* Willing to receive SMS
* Age ≥14 years
* Able to read and respond to text messages in English, Kiswahili or Luo, or have someone in the household who can help
* Receiving antenatal care at study facility
* Plan to be in the area for at least 3 months postpartum

Exclusion Criteria:

* participating in another study
* previously participated in this study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal Mortality | 28 days postpartum
  Death during 1st 28 days of life

SECONDARY OUTCOMES:
Cord care | 2-weeks postpartum
  Number of participants with no application of substances or chlorhexidine only to cord
Thermal Care | 24-hours postpartum
  Number of participants giving infant a bath in 1st 24 hours of life
Early Initiation of Breastfeeding | 1-hour postpartum
  Number of participants initiating breastfeeding in 1st hour of life
Appropriate Care-Seeking | 6-weeks postpartum
  Proportion of illness episodes with danger signs where the infant attended a medical facility
Maternal Knowledge of Neonatal Danger Signs | 6-weeks postpartum
  Number of danger signs or symptoms successfully named

OTHER OUTCOMES:
Home Visit Coverage | 2 years of study implementation
  Number of home visits performed by CHVs
Clinic Referrals | 2 years of study implementation
  Number of clinic referrals logged in dCHT by CHVs
Provider Workload | 2 years of study implementation
  Time on all CHV/supervisor duties
Acceptability | 2 years of study implementation
  Perception by CHVs that CHV-NEO is agreeable or satisfactory on the Acceptability of Intervention Measure (higher score is more acceptable)
Adoption | 2 years of study implementation
  Proportion of client messages replied to by CHV
Fidelity | 2 years of study implementation
  Number of client SMS responded to by CHV on time per SOP

CONTACTS AND LOCATIONS:
Overall Officials: Keshet Ronen, MPH, PhD, Principal Investigator — University of Washington; John Kinuthia, MBChB, MPH, Study Director — Kenyatta National Hospital
Locations (1):
- Kenyatta National Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data from CHV-NEO will be available at end of the project by contacting the study team at the University of Washington (chv-neo@uw.edu) or accessing data on GitHub.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the project.
Access Criteria: After publication of original data, data may be shared upon request with other investigators at academic, non-profit, or Kenyan government institutions in a limited data set. The final dataset will be stripped of identifiers prior to release for sharing. Investigators requesting access to data must sign a data-sharing agreement that provides for a commitment to: (1) using the data only for research purposes and not to identify any individual participant; (2) securing the data using appropriate computer technology; (3) not sharing the data with third parties, and (4) destroying or returning the data after analyses are completed. We reserve the right to limit data provided to outside investigators if we believe there is a possibility of deductive disclosure of subjects with unusual characteristics.

REFERENCES:
- [Derived] Ronen K, Pothan LC, Apondi V, Otieno FA, Mwakanema D, Otieno FO, Osborn L, Dettinger JC, Shrestha P, Manguerra H, Mukumbang F, Masinde M, Waweru E, Amulele M, Were C, Wasunna B, John-Stewart G, Weiner B, Means AR, Richardson BA, Hedstrom AB, Unger JA, Kinuthia J. Digital communication between mothers and community health workers to support neonatal health (CHV-NEO): study protocol for a randomized controlled trial. Trials. 2024 Oct 4;25(1):657. doi: 10.1186/s13063-024-08501-2. PMID 39367450